CLINICAL TRIAL: NCT00711737
Title: Open-label Study of the Changes in Metabolic Parameters in Patients Treated With Escitalopram for Six Months
Brief Title: Study of the Changes in Metabolic Parameters in Patients Treated With Escitalopram for Six Months
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Changi General Hospital, Changi General Hospital
Other Study IDs: 2008.06
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Major Depression; Generalized Anxiety Disorder; Panic Disorder
Keywords: metabolic parameters; escitalopram; metabolic syndrome; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Panic Disorder; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the changes in metabolic parameters in patients treated with escitalopram for six months for major depression, generalized anxiety disorder or panic disorder, with or without agoraphobia.

DETAILED DESCRIPTION:
This is an open-label study, with 4 scheduled visits. Recruitment of 100 subjects. Assessments include demographics, diagnosis, smoking frequency, Clinical Global Scale (CGI-S), weight, height,blood pressure, waist and hip circumference and fasting blood glucose and lipd profile.

Statistical analysis will be exploratory and mainly descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Give informed consent
* Requires pharmacological treatment with escitalopram for major depression, generalized anxiety disorder or panic disorder
* Aged 21 years old and above
* Able to comprehend and comply with protocol
* Not pregnant and if of child-bearing age, using adequate methods of contraception

Exclusion Criteria:

* Currently taking or has taken in previous 3 months, any other antidepressants, antipsychotics, mood stabilizers, weight loss or lipid-profile modifying drugs
* Contraindications to escitalopram
* Unstable medical illness and/or is already under treatment of diabetes, hypertension, dyslipidemia, ischemic heart disease
* History of non-response to escitalopram
* Meets IDF definition of metabolic syndrome
* Significant risk of suicide
* Primary diagnosis or comorbid diagnosis of psychotic disorder, bipolar disorder, substance dependence and/or dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients in psychiatric clinic in a general hosptial
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lai H Peh, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore